CLINICAL TRIAL: NCT00801138
Title: The Effect of Dexamethasone on the Duration of Interscalene Nerve Blocks With Ropivacaine or Bupivacaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A strong primary outcome crosses the efficacy boundary at the interim analysis
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-647
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia, Local; Shoulder Surgery
Keywords: ropivacaine; bupivacaine; glucocorticoid
MeSH Terms: interventions — Sodium Chloride; Dexamethasone; Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): Group 1 Ropivacaine: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline for interscalene block
  Interventions: Drug: saline; Drug: ropivacaine
- Group 2 (Placebo Comparator): Group 2 Bupivacaine: 30 ml 0.5% bupivacaine plus 2 ml 0.9% saline
  Interventions: Drug: saline; Drug: Bupivacaine
- Group 3 (Active Comparator): Group 3 Ropivacaine and dexamethasone: 30 ml 0.5% ropivacaine mixed with dexamethasone 8 mg (2 ml)
  Interventions: Drug: Dexamethasone; Drug: ropivacaine
- Group 4 (Active Comparator): Group 4 Bupivacaine and steroid: 30 ml 0.5% bupivacaine mixed with dexamethasone 8 mg (2 ml).
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine

INTERVENTIONS:
Drug: saline — 2 ml 0.9% saline (placebo)
  Arms: Group 1; Group 2
Drug: Dexamethasone — dexamethasone 8 mg (2 ml)
  Arms: Group 3; Group 4
Drug: ropivacaine — 30 ml 0.5% ropivacaine
  Arms: Group 1; Group 3
Drug: Bupivacaine — 30 ml 0.5% bupivacaine
  Arms: Group 2; Group 4

SUMMARY:
This study will test the hypothesis that adding dexamethasone significantly prolongs the duration of ropivacaine and bupivacaine analgesia, and that the magnitude of the effect differs among the two local anaesthetics.. Participants will be patients undergoing shoulder surgery with an interscalene nerve block.

DETAILED DESCRIPTION:
This is a double-blinded randomized study of four groups of patients undergoing shoulder surgery using interscalene nerve blocks. Participants will be randomized into one of four groups:

* Ropivacaine: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline (placebo) for interscalene block;
* Bupivacaine: 30 ml 0.5% bupivacaine plus 2 ml 0.9% saline (placebo);
* Ropivacaine and steroid: 30 ml 0.5% ropivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic;
* Bupivacaine and steroid: 30 ml 0.5% bupivacaine plus dexamethasone 8 mg (2 ml) mixed with the local anesthetic.

The primary outcome is the duration of the interscalene nerve block which is time to first analgesic request after PACU discharge.

Kaplan-Meier survival density estimation and stratified Cox proportional hazard regression were used to compare groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Patients undergoing shoulder procedures, such as rotator cuff repair, capsular shift, shoulder arthroplasty, subacromial decompression

Exclusion Criteria:

* Contraindications to interscalene block (Coagulopathy, infection at the needle insertion site, moderate to severe chronic obstructive pulmonary disease, contralateral pneumothorax or diaphragmatic paralysis)
* Pregnancy
* Pre-existing neuropathy involving the surgical limb
* Systemic glucocorticoid treatment (for 2 weeks or more) within six months of surgery
* Chronic opioid use (greater than 30 mg oral oxycodone equivalent per day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cummings, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; Ivan Parra Sanchez, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Group 1 Ropivacaine: 30 ml 0.5% ropivacaine plus 2 ml 0.9% saline for interscalene block
  Ropivacaine
  Placebo: saline
- Group 2: Group 2 Bupivacaine: 30 ml 0.5% bupivacaine plus 2 ml 0.9% saline
  Bupivacaine
  Placebo: saline
- Group 3: Group 3 Ropivacaine and dexamethasone:
  Ropivacaine plus dexamethasone
  Ropivacaine
  Dexamethasone: steroid
- Group 4: Group 4 Bupivacaine and steroid:
  Bupivacaine plus dexamethasone
  Bupivacaine
  Dexamethasone: steroid
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 54 | 56 | 54 | 54
Completed | 54 | 56 | 54 | 54
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 54 | 56 | 54 | 54 | 218
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 65] | 60 [51 to 68] | 59 [49 to 68] | 58 [53 to 64] | 58 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 21 | 22 | 83
  Male | 33 | 37 | 33 | 32 | 135

OUTCOME MEASURES:

1. Primary Outcome: The Duration of the Interscalene Nerve Block Which is Time to First Administration of Pain Medication After Block
Time Frame: Postoperative day 1, 2 and 3
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 56 | 54 | 54
hours | 11.8 [9.7 to 13.8] | 14.8 [11.8 to 18.1] | 22.2 [18.0 to 28.6] | 22.4 [20.5 to 29.3]

2. Secondary Outcome: Time to First Report of Pain
Time Frame: Postoperative day 1, 2 and 3
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 56 | 54 | 54
hours | 11.9 [9.2 to 13.8] | 14.7 [13.4 to 17.9] | 22.3 [18.0 to 27.2] | 25.7 [21.7 to 29.2]

3. Secondary Outcome: Median Maximum VAS Pain Scores at Rest
Description: Visual Analogue Scale (VAS) pain scale is used to describe the severity or intensity of pain. It ranges from 0 to 10. Zero indicates"no pain at all" and ten indicates "worst pain imaginable." , The higher of the score, the worse of the pain.
Time Frame: Postoperative day 1, 2 and 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 56 | 54 | 54
units on a scale | 5 [3 to 7] | 5 [3 to 7] | 4 [2 to 6] | 3 [0 to 5]

4. Secondary Outcome: Total Three-day Opioid Consumption in Oral Oxycodone Equivalent
Time Frame: Postoperative day 1, 2 and 3
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 54 | 56 | 54 | 54
milligrams | 75 [45 to 153] | 85 [51 to 118] | 79 [45 to 153] | 60 [47 to 105]

ADVERSE EVENTS:
Time Frame: 14 days after surgery
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/56 | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes